CLINICAL TRIAL: NCT02240680
Title: A 24 Week Randomized, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Trial of Once Daily Linagliptin, 5 Milligrams Orally, as Add on to Basal Insulin in Elderly Type 2 Diabetes Mellitus Patients With Insufficient Glycaemic Control
Brief Title: Linagliptin as Add on to Basal Insulin in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.149; 2014-000904-88 (EudraCT Number)
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- linagliptin 5 mg (Experimental): patient to receive a tablet of linagliptin 5 mg each day
  Interventions: Drug: linagliptin
- placebo (Placebo Comparator): patient to receive a tablet of placebo matching linagliptin 5 mg
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo matching linagliptin 5 mg
  Arms: placebo
Drug: linagliptin — 5 mg once a day
  Arms: linagliptin 5 mg

SUMMARY:
To investigate the efficacy, safety, and tolerability of linagliptin 5 milligrams once a day compared to placebo as as add-on therapy for 24 weeks to stable basal insulin treatment in elderly patients, 60 years of age and older, with Type 2 Diabetes Mellitus and insufficient glycaemic control.Stable background therapy of metformin and/or alpha-glucosidase inhibitors is also allowed.

In addition, this trial will assess if linagliptin reduces the risk of hypoglycaemia when added to background basal insulin therapy. The treatment duration of this trial (24 weeks) will enable assessment of the clinically relevant endpoint of a decrease in glycosylated Haemoglobin, a well-accepted measurement of chronic glycaemic control.

ELIGIBILITY:
Inclusion criteria:

* Patients must sign and date an Informed Consent consistent with International Conference on Harmonisation and Good Clinical Practice guidelines and local regulations prior to any evaluation and participation in the trial.
* Male and female patients with a clinical diagnosis of Type 2 Diabetes Mellitus, at the time of Informed Consent, who are:
* 60 years of age or older at informed consent or Screen Visit,
* taking stable doses of basal or biosimilar basal insulin [strictly inclusive of: insulin neutral protamine Hagedorn and isophane insulin; Humalog Basal (a suspension of insulin lispro protamine); insulin degludec; insulin detemir; and insulin glargine] for at least 4 weeks prior to randomisation (Visit 3) with dose adjustments up to a maximum of plus or minus 20% of baseline being allowed,
* may or may not be taking metformin immediate release or extended release [if the patient is taking metformin, stable dose must be maintained for at least twelve weeks without dose adjustments prior to randomisation (Visit 3)], and
* may or may not be taking alpha-glucosidase inhibitors [acarbose, miglitol, and voglibose; if the patient is taking alpha-glucosidase inhibitors, stable dose must be maintained for at least twelve weeks without dose adjustments prior to randomisation (Visit 3)].
* Patients must have an glycosylated Haemoglobin of 7.0% (53 millimoles per mole) to 10.0% (86 millimoles per mole) at the first visit (Screen).
* Patients must have a Body Mass Index of 45 kilogram/meter squared or less at the Screen Visit.
* In the investigator's opinion, patients must be reliable, compliant, and agree to cooperate with all planned future trial evaluations as explained in detail during the informed consent process and to be able to perform them.

Exclusion criteria:

* Impaired cognitive ability as supported by the Saint Louis University Mental Status Examination, additional assessment if necessary, and verified by the investigator at the Screen Visit.
* Depressed mood as supported by a score of 10 or more on the Patient Health Questionnaire at the Screen Visit.
* Type 1 Diabetes Mellitus as determined by past medical records and history.
* Acute coronary syndrome (non-ST Elevation Myocardial Infarction, ST Elevation Myocardial Infarction, and/or unstable angina pectoris), stroke or transient ischemic attack within 3 months prior to Screen Visit.
* Indication of liver disease determined during Screen and/or Run-In Period, defined by a serum level above 3 times the upper limit of normal in any of the following: alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase.
* Bariatric, gastric bypass, and other gastrointestinal procedures or surgeries (including all types of gastric banding, restriction, and/or LapBand) with the objective of promoting weight loss within the past two years at Screen Visit.
* Medical history of cancer (except for resected non-invasive basal or squamous cell carcinoma) and/or treatment for cancer within the last 5 years.
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells (malaria, babesiosis, haemolytic anaemia).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (145):
- United States (38):
  - Syed Research Consultants, LLC, Sheffield, Alabama
  - Precision Research Institute, LLC, Chula Vista, California
  - Aurora Care Clinic, LLC, Costa Mesa, California
  - Prime Care Clinical Research, Laguna Hills, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Internal Medicine of the Rockies, Colorado Springs, Colorado
  - Cohen Medical Research Associates, LLC, Delray Beach, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Clinical Research of Hollywood, Hollywood, Florida
  - East Coast Institute for Research LLC at NE FL Endo & Diabetes, Jacksonville, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Baptist Diabetes Associates, PA, Miami, Florida
  - International Research Associates, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - South Florida Research Solutions, LLC, Pembroke Pines, Florida
  - Georgia Clinical Research, LLC, Snellville, Georgia
  - Midwest Endocrinology, Crystal Lake, Illinois
  - American Health Network, Avon, Indiana
  - Accent Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - Clinical Research Associates of Central Pennsylvania, Altoona, Pennsylvania
  - Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Preferred Primary Care Phys, Uniontown, Pennsylvania
  - TLM Medical Services, LLC, Columbia, South Carolina
  - Advanced Research Associates, Hodges, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Arlington Family Research Center, Inc., Arlington, Texas
  - Renaissance Clinical Research and Hypertension of Texas, Dallas, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Science Advancing Medicine Clinical Research Center, San Antonio, Texas
  - Office of Dr. Val R. Hansen, Bountiful, Utah
  - Millennium Clinical Trials LLC, Arlington, Virginia
  - York Clinical Research, LLC, Norfolk, Virginia
  - Rowan Research, Inc., Spokane, Washington
  - Family Medical Clinic, Milwaukee, Wisconsin
- Australia (3):
  - AIM Centre, Merewether, New South Wales
  - Royal Brisbane & Women's Hospital-Endocrinology, Herston, Queensland
  - ECRU Maroondah, East Ringwood, Victoria
- Ham - PRAC Mortelmans, Oostham, Belgium
- Colombia (5):
  - CEQUIN, Armenia
  - Dexa Diabetes Servicios Médicos Ltda, Bogotá
  - CAFAM Caja de Compensación Familiar, Bogotá
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
  - Hospital Pablo Tobón Uribe, Medellín
- Denmark (8):
  - Aalborg Sygehus Syd, Aalborg
  - Sydvestjyst Sygehus Esbjerg, Endokrinologisk afdeling, Esbjerg
  - Frederiksberg Hospital, Endokrinologisk afd., Frederiksberg
  - Gentofte University Hospital, Hellerup
  - Kolding Sygehus, Kolding
  - Bispebjerg Hospital, København NV
  - Køge Sygehus, Køge
  - Roskilde Sygehus, Roskilde
- Finland (4):
  - Keravan terveyskeskus, Kerava
  - Terveystalo Oulu, Diapolis, Oulu
  - Lääkärikeskus Aava, Turku, Turku
  - TYKS, Turku
- Germany (6):
  - Gemeinschaftspraxis, Asslar, Aßlar
  - ikfe - Institut für klinische Forschung und Entwicklung Berlin GmbH, Berlin
  - Diabetologische Schwerpunktpraxis, Bosenheim, Bosenheim
  - Dünnwaldpraxis, Köln, Cologne
  - Praxis Dr. Naudts, Rodgau, Rodgau
  - Praxis Dr. Braun, Unterschneidheim, Unterschneidheim
- Greece (6):
  - "Korgialeneio-Benakeio" Hellenic Red Cross Hospital, Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General Hospital of Attiki "KAT-EKA", Kifissia
  - General Hospital of Nikaia, Nikaia
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Connolly Hospital Blanchardstown, Dublin, Ireland
- Japan (32):
  - Daishinkai Medical Corporation Ookuma Hospital, Aichi, Nagoya
  - Matsuyama Shimin Hospital, Ehime, Matsuyama
  - Iryohojin Kikuchi Naika Clinic, Gunma, Maebashi
  - Nakamura Digestive Organ Internal Medicine Clinic, Hokkaido, Bibai
  - Iida Medical Clinic, Hokkaido, Hakodate
  - Jiyugaoka Yamada Clinic, Hokkaido, Obihiro
  - Shinkotoni family Clinic, Hokkaido, Sapporo
  - Yoshida Memorial Hospital, Hokkaido, Sapporo
  - Teine Keijinkai Clinic, Hokkaido, Sapporo
  - Japan Community Health Care Organization Hokkaido Hospital, Hokkaido, Sapporo
  - Itabashi Diabetic medicine and Dermatology Clinic, Ibaraki, Koga
  - Nakakinen Clinic, Ibaraki, Naka
  - Takai Naika Clinic, Kanagawa, Kamakura
  - Kaneshiro DIAB Clinic, Kanagawa, I.M., Kanagawa, Sagamihara
  - Asahi Med. clinic, Kanagawa, I.M., Kanagawa, Yokohama
  - Ishikawa Med. Clinic, Kanagawa, I.M., Kanagawa, Yokohama
  - National Hospital Organization Yokohama Medical Center, Kanagawa, Yokohama
  - Okayama Saiseikai General Hospital Outpatient Center, Okayama, Okayama
  - AMC Nishi-umeda Clinic, Osaka, Osaka
  - Nissay Hospital Nippon Life Saiseikai Public Interest Incorporated Foundation, Osaka, Osaka
  - OCROM Clinic, Osaka, Suita
  - Saga Memorial Hospital, Saga, Saga
  - Asano Clinic, Saitama, Kawagoe
  - Hamamatsu Rosai Hospital, Shizuoka, Hamamatsu
  - Kuriyama Clinic, Tokyo, Adachi-ku
  - The Institute for Adult Deseases, Asahi Life Foundation, Tokyo, Chuo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Tokyo Center Clinic, Tokyo, Chuo-ku
  - AGE Makita Medical Clinic, Tokyo, Chuo-ku
  - Kobayashi Internal Medicine Clinic, Tokyo, Koto-ku
  - Kunitachi Naika Clinic, Tokyo, Kunitachi
  - Japanese Red Cross Medical Center, Tokyo, Shibuya-ku
- Mexico (6):
  - Investigación en Salud y Metabolismo S.C., Chihuahua City
  - Centro de At. e Inv.en Fact.de riesgo cardiovasc.Omega, S.C., México
  - Clinstile S.A. de C.V., México
  - CAIMED, México
  - CEDOPEC-Ctro Esp en Diab, Obesidad y Prev de Enf Cardiovasc, México
  - Asociación Mexicana para la Investigacion Clínica, A.C(AMIC), Pachuca
- New Zealand (3):
  - Middlemore Clinical Trials, Auckland
  - South Pacific Clinical Trials, Auckland, New Zealand
  - Christchurch Hospital, Christchurch
- Poland (3):
  - Medicome Sp. z o.o., Oświęcim
  - Omedica Centrum Medyczne, Poznan
  - NBR Polska, Warsaw
- Romania (3):
  - Nicodiab SRL, Bucharest, Bucharest
  - Pelican Impex SRL, Cabinet Nr. 15, Oradea
  - Mediab SRL, Târgu Mureş
- South Africa (9):
  - TREAD Research, Cape Town
  - Tiervlei Trial Centre, Cape Town
  - Paarl Research Centre, Cape Town
  - Soweto Clinical Trials Centre, Johannesburg
  - LCS Clinical Research Unit, Johannesburg
  - Resego Health Services, Johannesburg
  - Zinakekele Medical Centre, Kwamhlanga
  - Mzansi Ethical Research Centre, Middleburg
  - VX Pharma (Pty) Ltd Pretoria, Pretoria
- Spain (10):
  - Hospital A Coruña, A Coruña
  - Instituto de Ciencias Médicas, Alicante
  - Hospital Quiron. I.C.U., Barcelona
  - C.A.P. Sardenya, Barcelona
  - CAP Les Corts, Barcelona
  - CAP Canet de Mar, Canet de Mar
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Clínico de Valencia, Valencia
  - CAP El Remei, Vic
- United Kingdom (7):
  - The Haven Surgery, Burnhope
  - South Axholme Practice, Doncaster
  - Fowey Clinical Research Company Ltd, Fowey
  - Oak Tree Surgery, Liskeard
  - St. Mary's Hospital, Vectasearch Clinic, Newport, Newport
  - Mounts Bay Medical Ltd, Penzance
  - Rame Medical, Penntorr Health, Torpoint

REFERENCES:
- [Derived] Araki E, Unno Y, Tanaka Y, Sakamoto W, Miyamoto Y. Long-Term Efficacy and Safety of Linagliptin in a Japanese Population with Type 2 Diabetes Aged >/= 60 Years Treated with Basal Insulin: A Randomised Trial. Adv Ther. 2019 Oct;36(10):2697-2711. doi: 10.1007/s12325-019-01065-7. Epub 2019 Sep 3. PMID 31482511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was randomised, double blinded, placebo controlled, parallel study. Total 525 patients with type 2 diabetes mellitus (T2DM) and insufficient glycaemic control were screened. 302 patients were randomised into two groups. The trial was extended to 52 weeks for Japanese patients. 102 patients were identified and observed for the extended period.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that they (the subject) met all strictly implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Placebo (Up to 24 Weeks): Patients were orally administered with Placebo tablets (matching Linagliptin) once daily up to 24 weeks
- Linagliptin 5 Milligram (Up to 24 Weeks): Patients were orally administered with Linagliptin 5 milligram film-coated tablets once daily up to 24 weeks.
- Placebo (Up to 52 Weeks): Only Japanese patients were orally administered with Placebo tablets (matching Linagliptin) once daily up to 52 weeks
- Linagliptin 5 Milligram (Up to 52 Weeks): Only Japanese patients were orally administered with Linagliptin 5 milligram film-coated tablets once daily up to 52 weeks
Period: Overall Study (Up to 24 Weeks)
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks) | Placebo (Up to 52 Weeks) | Linagliptin 5 Milligram (Up to 52 Weeks)
Started | 151 | 151 | 0 | 0
Completed | 136 | 143 | 0 | 0
Not Completed | 15 | 8 | 0 | 0
Not completed — Adverse Event | 6 | 6 | 0 | 0
Not completed — Protocol Violation | 4 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — Other than specified | 1 | 0 | 0 | 0
Period: Japanese Patients (Up to 52 Weeks)
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks) | Placebo (Up to 52 Weeks) | Linagliptin 5 Milligram (Up to 52 Weeks)
Started | 0 | 0 | 50 | 52
Completed | 0 | 0 | 42 | 45
Not Completed | 0 | 0 | 8 | 7
Not completed — Adverse Event | 0 | 0 | 6 | 7
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): It includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks) | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data of age collected for all included patients in the study. Population: Treated set (TS): includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
  Years | 72.5 (5.6) | 72.3 (5.1) | 72.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Data of Gender collected of all patients included in the study. Population: Treated set (TS): includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
  Participants
    Female | 60 | 59 | 119
    Male | 91 | 92 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data for Ethnicity of patients collected under protocol for all included patients in the study. Population: Treated set (TS): includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
  Participants
    Hispanic or Latino | 19 | 15 | 34
    Not Hispanic or Latino | 132 | 136 | 268
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data for Race of patients collected under protocol for all included patients in the study. Population: Treated set (TS): It includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
  Participants
    American Indian or Alaska Native | 7 | 4 | 11
    Asian | 52 | 52 | 104
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 10 | 8 | 18
    White | 81 | 84 | 165
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1c (HbA1c) at baseline [Mean (Standard Deviation); unit: Percentage of HbA1c (%)] — HbA1c values measured at baseline in percent. HbA1c is a form of hemoglobin, a blood pigment that carries oxygen, which is bound to glucose. The term HbA1c also refers to glycated hemoglobin. High levels of HbA1c (Normal range is less than 6%) indicate poorer control of diabetes than level in normal range. Population: Full analysis set (FAS): Includes all patients randomised in the Treated Set who had a baseline and at least one on-treatment HbA1c value.
  Percentage of HbA1c (%)
    number analyzed (Participants) | 147 | 149 | 296
    (all) | 8.1 (0.7) | 8.2 (0.8) | 8.2 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) After 24 Weeks of Treatment.
Description: This outcome has measured difference between HbA1c values from baseline to 24 weeks post treatment. The term 'baseline' refers to the last observation prior to the administration of any randomised study medication. HbA1c is a form of hemoglobin, a blood pigment that carries oxygen, which is bound to glucose. The term HbA1c also refers to glycated hemoglobin. High levels of HbA1c (Normal range is less than 6%) indicate poorer control of diabetes than level in normal range.
Time Frame: Baseline and Week 24
Population: Full analysis set observed cases (FAS (OC)): Includes all patients randomised in the Treated Set who had a baseline and at least one on-treatment HbA1c value. These analyses used available data as observed while patients were on treatment. All values collected after a patient started rescue medication were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%) of HbA1c
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks)
Number analyzed (Participants) | 147 | 149
Percentage (%) of HbA1c | -0.38 (0.07) | -1.01 (0.06)
Statistical Analysis 1: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mixed model repeated measures(MMRM) included treatment, week and interaction as fixed effects, baseline HbA1c, daily basal insulin dose as covariates; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-0.81 to -0.46], Standard Error of Mean 0.09 — Adjusted mean of all differences between HbA1c at baseline and after 24 weeks. It is based on all patients in the model (not only patients with a baseline and week 24 measurement); MMRM including fixed effects treatment , week and treatment by week interaction linear covariates baseline HbA1c , baseline daily basal insulin and baseline HbA1c by week interaction and random effect for patient. Within-patient errors are modelled by unstructured covariance matrix. Adjusted mean is based on all patients in the model (not only patients with a baseline and week 24 measurement)

2. Secondary Outcome: Percentage of Patients Experiencing at Least One Hypoglycaemia Accompanied by a Prespecified Glucose Value.
Description: Hypoglycaemia accompanied by a prespecified glucose value is defined as any investigator reported hypoglycaemia (event or AE) with a reported blood glucose level of less than 54 milligram/deciLitre (3.0 millimole/Litre) or any investigator reported symptomatic hypoglycaemic AE with a reported blood glucose level of less or equal 70 milligram/deciLitre (3.9millimole/Litre) or any severe hypoglycaemic AE. Severe hypoglycaemia is an event that requires the assistance of another person to actively administer carbohydrates or glucagon because the patient is unable to take the substance on his or her own. The confidence intervals mentioned in measure of dispersion are exact 95% confidence interval by Clopper and Pearson. The percentage of patients with at least one hypoglycaemia accompanied by a glucose value less than 54mg/dL alone has also represented separately according American Diabetes Association definition of clinically significant hypoglycaemia.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients (%)
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks)
Number analyzed (Participants) | 147 | 149
Percentage of patients (%)
  Prespecified glucose value | 23.8 [17.2 to 31.5] | 30.9 [23.6 to 39.0]
  Glucose value <54 mg/dL | 15.0 [9.6 to 21.8] | 16.8 [11.2 to 23.8]
Statistical Analysis 1: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); For any hypoglycemia event accompanied by prespecified glucose value; Test type: Other; p = 0.1594, Regression, Logistic; A logistic regression model with treatment as fixed effect and baseline HbA1c and baseline daily basal insulin dose as linear covariates was applied; Odds Ratio (OR) = 1.464, 95% CI 2-sided [0.861 to 2.491], Standard Error of Mean 0.397 — The dispersion value standard error of the mean is actually standard error for odds ratio
Statistical Analysis 2: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); For glucose value < 54mg/dL according American Diabetes Association definition of clinically significant hypoglycaemia; Test type: Other; p = 0.6720, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.149, 95% CI 2-sided [0.604 to 2.188], Standard Error of Mean 0.377 — The dispersion value standard error of the mean is actually standard error for odds ratio

3. Secondary Outcome: Percentage of Patients With HbA1c<8.0%
Description: This is the percentage of patients with HbA1c on treatment <8.0% after 24 weeks of treatment. The confidence intervals mentioned in measure of dispersion are exact 95% CI by Clopper and Pearson.
Time Frame: 24 weeks
Population: Full analysis set (Non-completers considered failure)(FAS (NCF)): Includes all patients randomised in the Treated Set who had a baseline and at least one on-treatment HbA1c value. This analyses regarded missing values for binary efficacy endpoints as failure.
Measure: Number (95% Confidence Interval); unit: Percentage of patients (%)
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks)
Number analyzed (Participants) | 147 | 149
Percentage of patients (%) | 40.2 [29.9 to 51.3] | 70.1 [59.4 to 79.5]
Statistical Analysis 1: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); Test type: Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.018, 95% CI 2-sided [2.468 to 10.206], Standard Error of Mean 1.818 — The dispersion value standard error of the mean is actually standard error of odds ratio

4. Secondary Outcome: Percentage of Patients With HbA1c on Treatment <7.0%
Description: This is the percentage of patients with HbA1c on treatment <7.0% after 24 weeks of treatment. The confidence intervals mentioned in measure of dispersion are exact 95% CI by Clopper and Pearson.
Time Frame: 24 weeks
Population: Full analysis set non-completers considered failure (FAS (NCF)): Includes all patients randomised in the treated set who had a baseline and at least one on-treatment HbA1c value. This analyses regarded missing values for binary efficacy endpoints as failure.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients (%)
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks)
Number analyzed (Participants) | 147 | 149
Percentage of Patients (%) | 14.6 [9.3 to 21.4] | 37.8 [29.8 to 46.2]
Statistical Analysis 1: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); Test type: Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.689, 95% CI 2-sided [2.485 to 8.848], Standard Error of Mean 1.519 — The dispersion value standard error of the mean is actually standard error of odds ratio

5. Secondary Outcome: Percentage of Patients With HbA1c Lowering by at Least 0.5%.
Description: The percentage of patients who attained lowering of HbA1c by ≥0.5% from baseline after 24 weeks of treatment were analysed. The confidence intervals mentioned in measure of dispersion are exact 95% CI by Clopper and Pearson.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of patients (%)
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks)
Number analyzed (Participants) | 147 | 149
Percentage of patients (%) | 37.4 [29.6 to 45.8] | 69.1 [61.0 to 76.4]
Statistical Analysis 1: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); Test type: Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 3.731, 95% CI 2-sided [2.302 to 6.048], Standard Error of Mean 0.920 — The dispersion value standard error of the mean is actually standard error of odds ratio

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: This outcome has measured difference between FPG values from baseline to 24 weeks post treatment. The term 'baseline' refers to the last observation prior to the administration of any randomised study medication
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram/decilitre
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 Milligram (Up to 24 Weeks)
Number analyzed (Participants) | 147 | 149
milligram/decilitre | 0.2 (3.6) | -11.3 (3.3)
Statistical Analysis 1: Comparison: Placebo (Up to 24 Weeks) vs Linagliptin 5 Milligram (Up to 24 Weeks); Test type: Superiority; p = 0.0178, Mixed Models Analysis; Mixed model repeated measures(MMRM) included treatment, week and interaction as fixed effects, baseline HbA1c, FPG, daily insulin dose as covariates; Mean Difference (Final Values) = -11.5, 95% CI 2-sided [-21.0 to -2.0], Standard Error of Mean 4.8 — [estimate comment as in outcome 1, analysis 1]; MMRM including fixed effects treatment, week and treatment by week interaction, linear covariates baseline HbA1c, baseline daily basal insulin, baseline FPG and baseline FPG by week interaction and random effect for patient. Within-patient errors are modelled by unstructured covariance matrix. Adjusted mean is based on all patients in the model (not only patients with a baseline and week 24 measurement)

ADVERSE EVENTS:
Time Frame: The adverse events were reported by overall population from first drug administration up to treatment period of 24 weeks, until 7 days after last drug administration. The adverse events were reported by Japanese population from first drug administration up to treatment period of 52 weeks, until 7 days after last drug administration.
Description: An AE was defined as any untoward medical occurrence, including an exacerbation of a preexisting condition, in a patient in a clinical investigation who received a pharmaceutical product. A treated set (TS) was used for analysis of adverse events. TS includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Linagliptin 5 mg (Up to 24 Weeks): Patients were orally administered with Linagliptin 5 mg film-coated tablets once daily up to 24 weeks.
- Placebo (Up to 52 Weeks): Japanese patients were orally administered with Placebo tablets (matching Linagliptin) once daily up to 52 weeks
- Linagliptin 5mg (Up to 52 Weeks): Japanese patients were orally administered with Linagliptin 5 mg film-coated tablets once daily up to 52 weeks.
Arm/Group | Placebo (Up to 24 Weeks) | Linagliptin 5 mg (Up to 24 Weeks) | Placebo (Up to 52 Weeks) | Linagliptin 5mg (Up to 52 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/151 | 2/151 | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 21/151 | 19/151 | 7/50 | 13/52
Other Adverse Events (participants affected / at risk) | 58/151 | 72/151 | 19/50 | 37/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Up to 24 Weeks) (N=151) | Linagliptin 5 mg (Up to 24 Weeks) (N=151) | Placebo (Up to 52 Weeks) (N=50) | Linagliptin 5mg (Up to 52 Weeks) (N=52)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 2
Diabetic retinopathy (Eye disorders) | 0 | 2 | 0 | 2
Glaucoma (Eye disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 1 | 1 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Up to 24 Weeks) (N=151) | Linagliptin 5 mg (Up to 24 Weeks) (N=151) | Placebo (Up to 52 Weeks) (N=50) | Linagliptin 5mg (Up to 52 Weeks) (N=52)
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Large intestine polyp (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Bronchitis (Infections and infestations) | 4 | 7 | 0 | 5
Urinary tract infection (Infections and infestations) | 9 | 10 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 8 | 11 | 3 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 38 | 51 | 14 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 3 | 0 | 3

LIMITATIONS AND CAVEATS:
For patients in Japan, a local protocol amendment was introduced, and according to it the study was extended to 52 weeks for Japanese population only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT02240680/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02240680/SAP_001.pdf